CLINICAL TRIAL: NCT03691870
Title: Transvenous Approach for the Treatment of Cerebral Arteriovenous Malformations (TATAM): A Randomized Controlled Trial and Registry
Brief Title: Transvenous Approach for the Treatment of Cerebral Arteriovenous Malformations
Acronym: TATAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18.118
Record Dates: First submitted 2018-09-20; First posted 2018-10-02 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Arteriovenous Malformations, Cerebral; Unruptured Brain Arteriovenous Malformation; Ruptured Brain Arteriovenous Malformation
Keywords: brain arteriovenous malformation; Arteriovenous malformations; AVM; BAVM; stroke; intracranial hemorrhage; congenital abnormalities; aneurysm; vascular malformations; cardiovascular abnormalities; cardiovascular diseases; vascular diseases
MeSH Terms: conditions — Intracranial Arteriovenous Malformations; Arteriovenous Malformations; Stroke; Intracranial Hemorrhages; Congenital Abnormalities; Aneurysm; Vascular Malformations; Cardiovascular Abnormalities; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard Trans-Arterial Embolization (TAE) (Active Comparator): The standard TAE, without TVE, is used in patient allocated standard treatment.
  The arterial approach will consist of at least one attempted catheterization for trans-arterial injection of liquid embolic.
  Patients incompletely treated at the time of the final embolization procedure are adjudicated a failure to reach the primary outcome and can be treated using alternative standard options (including surgery, radiation therapy, conservative management). In addition, patients of the control group can also be offered TVE, if still feasible, once the TAE has been adjudicated to be a failure.
  If the operator deems, on the table, for a trans-arterial injection to be too dangerous, no arterial injection is necessary. Treatment, where indicated, can be completed through other means.
  Interventions: Procedure: Standard Trans-Arterial Embolization (TAE)
- Trans-Venous Embolization (TVE) (+/- Arterial) strategy (Experimental): The experimental treatment is an attempt to completely occlude the AVM using venous catheterization and retrograde EVOH injection during the final session. TAE can be performed to prepare for final TVE during the same or one previous preparatory session, or TAE can be used to rescue an incomplete TVE. In some patients, balloon catheterization is used trans-arterially to assist TVE.
  It will be permissible to perform more than one treatment session when deemed necessary (occasionally to treat an AVM through the trans-venous route requires a two-stage approach, with a single trans-arterial attempt to decrease AVM filling prior to the definitive trans-venous approach, and this will be permitted).
  The trans-venous strategy will consist of at least one transvenous injection of ethyl vinyl alcohol (EVOH), with the choice of delivery microcatheters and other technical details left to the individual operator's discretion).
  Interventions: Procedure: Trans-Venous Embolization (TVE)

INTERVENTIONS:
Procedure: Standard Trans-Arterial Embolization (TAE) — The standard TAE, without TVE, is used in patient allocated standard treatment. The arterial approach will consist of at least one attempted catheterization for trans-arterial injection of liquid embolic.
  If the operator deems, on the table, for a trans-arterial injection to be too dangerous, no arterial injection is necessary. Treatment, where indicated, can be completed through other means.
  Arms: standard Trans-Arterial Embolization (TAE)
Procedure: Trans-Venous Embolization (TVE) — The experimental treatment is an attempt to completely occlude the AVM using venous catheterization and retrograde EVOH injection during the final session.
  The trans-venous strategy will consist of at least one transvenous injection of ethyl vinyl alcohol (EVOH), with the choice of delivery microcatheters and other technical details left to the individual operator's discretion.
  Arms: Trans-Venous Embolization (TVE) (+/- Arterial) strategy

SUMMARY:
A new endovascular route for the treatment of brain AVMs may be possible in some cases: Trans-Venous Embolization (TVE). The technique uses microcatheters to navigate to the draining veins of AVM, to reach and then fill the AVM nidus retrogradely with liquid embolic agents until the lesion is occluded. This technique has the potential to improve on some of the problems with the arterial approach to AVM embolization, such as a low overall occlusion rate. However, by occluding the vein first, and filling the lesion with the embolic agent in a retrograde fashion, the method transgresses a widely held dogma in the surgical or endovascular treatment of AVMs: to preserve the draining vein until all afferent vessels have been occluded. Nevertheless, the initial case series have shown promising results, with high occlusion rates, and few technical complications.

The method is increasingly used in an increasing number of centers, but there is currently no research protocol to guide the use of this promising but still experimental treatment in a prudent fashion. Care trials can be designed to offer such an experimental treatment, taking into account the best medical interests of patients, in the presence of rapidly evolving indications and techniques.

ELIGIBILITY:
Inclusion Criteria:

* Any patient harboring a brain AVM (ruptured or unruptured) in whom TVE is considered a promising but yet unproven therapeutic option by the participating clinicians can be submitted to the Case Selection Committee.
* Patients must be in stable, non-urgent clinical condition, with the acute phase of the AVM rupture resolved (where applicable).
* Case must be approved by the CSC.

Notes on potentially suitable cases:

1. Current indications may include (but are NOT restricted to) brain AVMs with a small <3 cm nidus (or small residual nidus), with a single draining vein, and for which curative treatment can be attained with one or at most two treatment sessions.
2. Physicians are not required to submit cases prior to any or all treatment; a case can be submitted to the CSC for consideration after previous treatments (including previous arterial embolization sessions) have been performed. The timing of the submission of the case will be left to individual operators. Previously treated AVMs (by any other modality: embolization/surgical resection/radiosurgery) are not excluded from TATAM.

Exclusion Criteria:

* Absolute contra-indication to endovascular treatment or anesthesia.
* Inability to obtain informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Angiographic evidence of residual AVM at time of confirmatory catheter angiography. | 3 months +/- 1 month following embolization
  Angiographic evidence of residual AVM at time of confirmatory catheter angiography

SECONDARY OUTCOMES:
Failure to safely and effectively position the embolization microcatheter. | within day of procedure
  Failure to reach a safe and effective microcatheter position for embolization.
Any procedural complication leading to transient new neurological deficit. | <5 days
  Any procedural complication leading to transient new neurological deficit.
Any procedural complication leading to new neurological deficit. | ≥5 days
  Any procedural complication leading to new neurological deficit.
Any treatment-related complication that prolongs hospitalization by ≥5 days. | Within one week
  Any treatment-related complication that prolongs hospitalization by ≥5 days.
Incidence of new ischemia following treatment (Brain MR imaging prior to discharge with diffusion sequences). | within 5 days post procedure
  Incidence of new ischemia following treatment (Brain MR imaging prior to discharge with diffusion sequences).
Length of hospitalization (days). | ≥5 days
  Length of hospitalization (days).
Patient discharge to a location that is not his/her home. | through to 3 (+/- 1) months follow-up
  Discharge to location other than home.
mRS at discharge and 3(+/-1) months. | through to 3 (+/- 1) months follow-up
  mRS at discharge and 3(+/-1) months.
Incidence of new admission to hospital during follow-up. | Within 3 +/- months post final treatment
  Incidence of new admission to hospital during follow-up.
Incidence of intracranial hemorrhage during follow-up. | Within 3 +/- months post final treatment
  Incidence of intracranial hemorrhage during follow-up.
Incidence of residual AVM on confirmatory catheter angiography at 3(+/-1) months post-treatment. | at 3(+/-1) months post-treatment.
  Incidence of residual AVM on confirmatory catheter angiography at 3(+/-1) months post-treatment.

CONTACTS AND LOCATIONS:
Locations (9):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
- France (7):
  - Centre hospitalier universitaire de Bordeaux, Bordeaux
  - Centre hospitalier régional universitaire de Brest, Brest
  - Centre hospitalier universitaire de Grenoble, Grenoble
  - Centre hospitalier universitaire Limoges, Limoges
  - Hôpital Forndation Adolphe de Rothschild, Paris
  - Centre hospitalier universitaire de Rouen Normandie, Rouen
  - Centre hospitalier universitaire de la Réunion, Saint-Paul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Beijnum J, van der Worp HB, Buis DR, Al-Shahi Salman R, Kappelle LJ, Rinkel GJ, van der Sprenkel JW, Vandertop WP, Algra A, Klijn CJ. Treatment of brain arteriovenous malformations: a systematic review and meta-analysis. JAMA. 2011 Nov 9;306(18):2011-9. doi: 10.1001/jama.2011.1632. PMID 22068993
- [Background] Iosif C, Mendes GA, Saleme S, Ponomarjova S, Silveira EP, Caire F, Mounayer C. Endovascular transvenous cure for ruptured brain arteriovenous malformations in complex cases with high Spetzler-Martin grades. J Neurosurg. 2015 May;122(5):1229-38. doi: 10.3171/2014.9.JNS141714. Epub 2015 Mar 20. PMID 25794338
- [Background] Kessler I, Riva R, Ruggiero M, Manisor M, Al-Khawaldeh M, Mounayer C. Successful transvenous embolization of brain arteriovenous malformations using Onyx in five consecutive patients. Neurosurgery. 2011 Jul;69(1):184-93; discussion 193. doi: 10.1227/NEU.0b013e318212bb34. PMID 21346657
- [Background] Mendes GAC, Kalani MYS, Iosif C, Lucena AF, Carvalho R, Saleme S, Mounayer C. Transvenous Curative Embolization of Cerebral Arteriovenous Malformations: A Prospective Cohort Study. Neurosurgery. 2018 Nov 1;83(5):957-964. doi: 10.1093/neuros/nyx581. PMID 29281075
- [Background] Zhang G, Zhu S, Wu P, Xu S, Shi H. The transvenous pressure cooker technique: A treatment for brain arteriovenous malformations. Interv Neuroradiol. 2017 Apr;23(2):194-199. doi: 10.1177/1591019916682357. Epub 2016 Dec 5. PMID 27913800
- [Background] Raymond J, Darsaut TE, Altman DG. Pragmatic trials can be designed as optimal medical care: principles and methods of care trials. J Clin Epidemiol. 2014 Oct;67(10):1150-6. doi: 10.1016/j.jclinepi.2014.04.010. Epub 2014 Jul 16. PMID 25042688
- [Background] Raymond J, Fahed R, Darsaut TE. Randomize the first patient. J Neuroradiol. 2017 Sep;44(5):291-294. doi: 10.1016/j.neurad.2017.03.004. Epub 2017 May 3. No abstract available. PMID 28478113
- [Derived] Raymond J, Darsaut TE, Saleme S, Rouchaud A, Iancu D, Roy D, Weill A, Olijnyk L, Jabre R, Bojanowski MW, Chaalala C, Roberge D, Boubagra K, Heck O, Rempel JL, Papagiannaki C, Barreau X, Marnat G, Gentric JC, Ognard J, Nico L, Bintner M, Gauthier Lasalarie P, Veyrieres JB, Piotin M, Escalard S, Pereira VM, Abud DG, Zehr J, Chagnon M, Nguyen TN, Mathieu D, Gevry G, Klink R, Lorian E, Mounayer C; TATAM Collaborative Group. Transvenous Approach for the Treatment of Cerebral Arteriovenous Malformations: A Randomized Comparison With Transarterial Embolization. Stroke. 2025 Jun;56(6):1396-1403. doi: 10.1161/STROKEAHA.124.049109. Epub 2025 Mar 27. PMID 40143818
- [Derived] Fahed R, Darsaut TE, Mounayer C, Chapot R, Piotin M, Blanc R, Mendes Pereira V, Abud DG, Iancu D, Weill A, Roy D, Nico L, Nolet S, Gevry G, Raymond J. Transvenous Approach for the Treatment of cerebral Arteriovenous Malformations (TATAM): Study protocol of a randomised controlled trial. Interv Neuroradiol. 2019 Jun;25(3):305-309. doi: 10.1177/1591019918821738. Epub 2019 Feb 4. PMID 30843441